CLINICAL TRIAL: NCT02172638
Title: Ensayo clínico Comparando Recuperación Postoperatoria Tras Protocolo FAST- TRACK Vs. Manejo Clásico en Cáncer de Ovario Avanzado
Brief Title: Postoperatory Recovery in Advanced Ovarian Cancer, Fast-Track Protocol vs. Classical Management
Acronym: PROFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR(AMI)136/2014
Record Dates: First submitted 2014-06-13; First posted 2014-06-24 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Median Length of Stay; Readmission Rate; Surgery Related Complications Rate; Cost Per Patient Rate
Keywords: Enhanced Recovery After Surgery; ERAS; Fast-Track; Ovarian cancer; Gynecologic surgery; Gynecology oncology; Median length of stay; Readmission rate; Surgery related complications; Cost
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Enhanced Recovery After Surgery

ARMS (2):
- FAST-TRACK Group (Experimental): Patients in this group will be managed according to an specifically designed FAST-TRACK protocol which will include: Preoperatory nutritional management and coaching by surgeon, anesthetist, nutritionist and specifically trained nurse personnel, reduced preoperatory fasting, avoiding use of intraabdominal drainages, specific anesthetic management to reduce intraoperative stress, avoiding use of Nasogastric tube, avoiding the need for major opioid in postoperatory analgesia and use of an standardized postoperatory management protocol directed to obtain an early oral intake and mobilization with a the goal of normal diet and deambulation in the 3rd day after surgery.
  Interventions: Procedure: Fast-Track Protocol
- Classical management group (Active Comparator): Patients assigned to this group will receive the standard management preformed in our center until now. This management includes a preoperatory control exclusively by the surgeon and anesthetist, minimum of 8h fasting previous to surgery, loose use of intraabdominal drainage , systematic use of nasogastric tube whenever rectum resection or omentectomy is performed, Postoperative analgesia following standing Vall d'Hebron protocols for Moderate-severe postoperative pain, which include use of combined analgesia with non opioids drugs and major Opioids, and usual flexible, non standardized postoperatory management with mobilization and oral intake progression depending on perceived evolution by attending surgeon.
  Interventions: Procedure: Usual management

INTERVENTIONS:
Procedure: Fast-Track Protocol
  Other Names: Enhanced Recovery After Surgery; ERAS protocol
  Arms: FAST-TRACK Group
Procedure: Usual management
  Other Names: Classical management; Conventional care
  Arms: Classical management group

SUMMARY:
The concept of Fast-trak or Enhanced Recovery After Surgery ( ERAS) represents a new approach to the management of patients undergoing major surgery that re-examine traditional practices, replacing them if necessary with the best evidence based practices, creating a multimodal perioperative care pathway designed to achieve early recovery. In Colorectal Cancer Surgery , as well as in a number of other procedures it has been shown to reduce Hospitalization by more than 30% without increasing the rate complications or readmissions.

However information on the results of Fast-track protocols when applied to Gynecological patients is sparse, being especially notorious the lack of data regarding the efficacy of Fast-track in the management of Advanced Gynecological cancer.

Hypothesis: the application of a Fast-Track protocol in the management of patients with advanced Ovarian Cancer( Stage III, IV and relapses) may improve the postoperatory recovery of these patients allowing for an early discharge and significant cost reduction, when compared with de usual management, without increasing the number readmission or surgery related complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more
* Advanced ovarian cancer ( FIGO Stages III-IV, and relapses) tributary to laparotomic surgical management.
* Patient accepts participation in the study and signs informed consent.

Exclusion Criteria:

* ASA IV
* Active ischemic cardiac condition
* Advanced cirrhosis ( Child-Pugh B -C).
* Severe Psychiatric condition ( patient not capable of giving her informed consent properly, not capable or not willing to attend Follow-up visits).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
median length of stay | participants will be followed for the duration of hospital stay, an expected average of 2 weeks.

SECONDARY OUTCOMES:
Number of readmissions related to postoperative complications. | 28 days after surgery
  To determine if there is an statistically significant difference in the readmission rate related to postoperative complications between the Fast-track and Classical management groups.
Number of surgery related complications | 28 days after surgery.
  To determine if there is an statistically significant difference in surgery related complications rates between the Fast-track and Classical management groups.
  The number and severity will be recorded. as graded in the Clavien-Dindo Classification of Surgical Complications.
Cost per patient | 28 days after surgery
  To determine if the application of a Fast-Track protocol in advanced ovarian cancer patients generates a significant cost per patient reduction when compared with classical management. The total cost for Hospitalization , readmissions and surgery related complications will be assessed according to the Public prices published in : SLT/383/2009, 21th January "Diari Oficial de la Generalitat de Catalunya" Núm. 5325 - 24.2.2009.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil Moreno, MD, Study Director — Hospital Vall d'Hebron; José Luis Sánchez Iglesias, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Delaney CP, Fazio VW, Senagore AJ, Robinson B, Halverson AL, Remzi FH. 'Fast track' postoperative management protocol for patients with high co-morbidity undergoing complex abdominal and pelvic colorectal surgery. Br J Surg. 2001 Nov;88(11):1533-8. doi: 10.1046/j.0007-1323.2001.01905.x. PMID 11683754
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396
- [Derived] Sanchez-Iglesias JL, Carbonell-Socias M, Perez-Benavente MA, Monreal Clua S, Manrique-Munoz S, Garcia Gorriz M, Burgos-Pelaez R, Segurola Gurrutxaga H, Pamies Serrano M, Pilar Gutierrez-Barcelo MD, Serrano-Castro S, Balcells-Farre MT, Perez-Barragan C, Scaillet-Houberechts A, Cossio-Gil Y, Gil-Moreno A. PROFAST: A randomised trial implementing enhanced recovery after surgery for highcomplexity advanced ovarian cancer surgery. Eur J Cancer. 2020 Sep;136:149-158. doi: 10.1016/j.ejca.2020.06.011. Epub 2020 Jul 18. PMID 32688208
- See also: Related Info — http://www.erassociety.org/